CLINICAL TRIAL: NCT02818985
Title: Intra-articular Dexamethasone vs Intra-articular Dexamedetomidine
Brief Title: Analgesia in Knee Arthroscopic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM2016
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexamethasone (Active Comparator): patients will receive intra-articular 8 mg dexamethasone added to 18 mL 0.25% bupivacaine into the knee joint.
  Interventions: Drug: Dexamethasone
- Dexmedetomidine (Active Comparator): patients will receive intra-articular 1ug/kg dexmedetomidine added to 18 mL 0.25% bupivacaine into the knee joint.
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): patients will receive intra-articular 18 mL 0.25% bupivacaine and 2mL isotonic saline into the knee joint.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — patients will receive intra-articular 8 mg dexamethasone added to 18 mL 0.25% bupivacaine into the knee joint.
  Arms: Dexamethasone
Drug: Dexmedetomidine — patients will receive intra-articular 1ug/kg dexmedetomidine added to 18 mL 0.25% bupivacaine into the knee joint.
  Arms: Dexmedetomidine
Drug: Saline — patients will receive intra-articular 18 mL 0.25% bupivacaine and 2mL isotonic saline into the knee joint.
  Arms: Control

SUMMARY:
Pain relief in knee Arthroscopic Surgery is essential for rapid recovery of function.

DETAILED DESCRIPTION:
Intra-articular analgesia is useful in reducing patients' postoperative disability. It anticipates and prevents the onset of pain, and helps avoid the need for additional drugs. Usually it is possible to reach good analgesia in the immediate postoperative period by the administration of analgesic drugs. Recently, intra-articular administration of different anaesthetic substances with a local action (e.g. bupivacaine) has been introduced in clinical practice. The aim of the administration of these substances should not be the reduction of postoperative pain, but its prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for knee arthroscopy under spinal anaesthesia

Exclusion Criteria:

* Diabetes Mellitus
* Contraindication to spinal anesthesia
* Patient refusal

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
pain free time | 48 hours
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut Univerisity
Locations (1):
- Seham Mohamed Moeen Ibrahim, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Moeen SM, Ramadan IK, Elkady HA. Dexamethasone and Dexmedetomidine as an Adjuvant to Intraarticular Bupivacaine for Postoperative Pain Relief in Knee Arthroscopic Surgery: A Randomized Trial. Pain Physician. 2017 Nov;20(7):671-680. PMID 29149146